CLINICAL TRIAL: NCT03692377
Title: How Young is Too Young for Virtual Reality ? Determination of the Usability and Acceptability of Virtual Reality for Health Care Purposes Among Children 2-6 Years of Age in the Emergency Department
Brief Title: How Young is Too Young for Virtual Reality? Determining Usability and Acceptability in Ages 2-6 in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ran Goldman, Professor and Co-head of the Division of Clinical Pharmacology, Division of Emergency Medicine, Department of Pediatrics; Investigator, BC Children's Hospital, University of British Columbia
Other Study IDs: H18-01924
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Child, Preschool
Keywords: Virtual Reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children Aged 2-6: Children 2 to 6 years of age who are arriving with a guardian to the Emergency Department with a low acuity condition (Canadian Triage scale (CTAS) 4 or 5) and are waiting to be seen by the doctor, or are waiting for test results.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Stage 1 : Demonstration of the use of the VR headset by the research assistant (anticipated 1-2 min) Stage 2 : Child will choose the application they would like to see - they will be shown 3 pages of the three applications offered - see Fig 1 (anticipated 1-2 min) Stage 3 : Handling of the VR headset by the child (anticipated 1 min) Stage 4 : Applying the headset on the eyes of the child with software application (anticipated 1 min) Stage 5 : The child use the VR set and application (up to 10 minutes) Stage 6 : Removal of the headset (anticipated 1 min) Stage 7 : Questionnaire to child (interview - 2 minutes) Stage 8 : Questionnaire to parents/guardians (interview - 2 minutes)

SUMMARY:
Children who present to the emergency department often require painful procedures (intravenous catheterization, laceration repair, fracture reduction, etc.). Virtual reality (VR) has been presented as a way of managing pain and anxiety in children undergoing painful procedures but most studies are limited to children 6 or older. The present study seeks to determine the youngest age (2-6) of future subjects in research of VR and clinical care.

Virtual Reality is an immersive experience using sight, sound, and position sense. Using VR may enhance distraction during the painful procedure and may reduce attention to pain.

Investigators will instruct and observe children age 2-6 in using a VR device and document how easy the device is to use for the child. The children will have the opportunity to select an application and play with the device for 10 minutes before being asked about their experience with the device. Parents/Guardians will also be asked about their child's experience with the device.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 2-6 years of age
2. Patients arrived with a legal guardian to the emergency department
3. Parents will sign a consent form and children will agree verbally to participate
4. Triage category 4 or 5 (lowest acuity)

Exclusion Criteria:

1. Children with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay, autism, neurological or other condition limiting communication)
2. Facial features or injury prohibiting wearing the VR goggles
3. Painful procedures in the emergency before being approached (such as blood testing, IV, catheterization, immunization, laceration repair)
4. Child is suffering pain or distress at a level that prohibit focusing on the study for 20 minutes, as assessed by the research assistant

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 2 to 6 years of age who are arriving with a guardian to the Emergency Department with a low acuity condition (Canadian Triage scale (CTAS) 4 or 5) and are waiting to be seen by the doctor, or are waiting for test results.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-09-21 (Estimated); Study Completion 2019-09-21 (Estimated)

PRIMARY OUTCOMES:
Usability in Stage 4 (Applying the headset on the eyes of the child with software application) as measured by a five point scale. | Recorded during Stage 4 of the procedure
  The research assistant will assess how the child reacts to wearing VR as measured by a five point scale:
  1. - Child tries to use the headset themselves with no help
  2. - Child helps the research assistant to put the headset on their face
  3. - Child is passive while the research assistant to put the headset on their face
  4. - Child resist by pushing the research assistant's hands
  5. - Child significantly resist/ cry/ wave arms / push feet

SECONDARY OUTCOMES:
Time of demonstration required by child measured in seconds | Recorded during Stage 1 of intervention, before child puts headset on. Up to 120 seconds.
  Length of Time (seconds) the demonstration took until the child was ready to wear the VR headset
Mood/Behaviors during Handling of VR rated 1-100 on a Visual analogue scale | Recorded during Stage 3 of intervention. Up to 1 minute while child handles and puts on headset.
  Rated 1-100 on a Visual analogue scale from extremely negative to extremely positive by the research assistant.
Time using VR in minutes | Recorded during Stage 5 of the procedure. Up to 10 minutes.
  Length of Time (Minutes) the child was using the VR set on their head (up to 10 minutes)
Willingness to Return VR as measured by a three point scale | Recorded during Stage 6 of the procedure
  The research assistant will record willingness to return VR as measured by a three point scale:
  1. - Give away the headset after requested to do so once
  2. - Give away the headset after requested to do so several times
  3. - Want to continue playing and does not give the set away
Patient experience questions as measured by a 4 point scale and open ended question | Immediately after the intervention (within 10 minutes)
  The research assistant will ask the patient four questions on a four point scale:
  How easy or hard it was to wear the VR goggles [1-very hard …………. 4-very easy] How easy or hard it was to see the video [1-very hard …………. 4-very easy] Do they want their parents to also try the VR goggles [1-not at all …………. 4-yes, immediately] Would they like to play again with the VR goggles [1-not at all …………. 4-yes, immediately]
  One open ended question will be asked about any problems with VR.
Parent experience questions as measured by a 4 point scale and open ended question | Immediately after the intervention (within 10 minutes)
  The research assistant will ask the patient two questions on a four point scale:
  How easy or hard it was for your child to wear the VR goggles [1-very hard …………. 4-very easy] Do they want their child to try the VR goggles next time they need a procedure in the hospital
  [1-not at all …………. 4-yes, immediately]
  One open ended question will be asked about any problems with VR.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Goldman, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada